CLINICAL TRIAL: NCT02914717
Title: One Year Outcome of Golimumab for Patients With Moderate-to-severe Ulcerative Colitis: a Retrospective Multi-centre Belgian Cohort Study
Brief Title: The Belgian SMART Study Evaluating the Use of Golimumab for Ulcerative Colitis
Acronym: BE SMART
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW (Other); Imelda Hospital, Bonheiden (Other); AZ Delta (Other); University Hospital, Ghent (Other); University Hospital, Antwerp (Other); Ziekenhuis Oost-Limburg (Other); Onze Lieve Vrouw Hospital (Other); General Hospital Groeninge (Other); University of Liege (Other); Clinique Saint Joseph, Liège (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Erasme University Hospital (Other); Chwapi Tournai (Unknown); AZ Jan Palfijn Gent (Other); CHR Verviers (Unknown); Virga Jesse Hasselt (Unknown); Damiaanziekenhuis Oostende (Unknown); AZ Sint-Lucas Brugge (Other)
Responsible Party: Sponsor
Other Study IDs: S59335
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2017-10

CONDITIONS: Ulcerative Colitis
Keywords: golimumab
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory condition causing continuous mucosal inflammation of the colon, which is accompanied by episodes of bloody diarrhoea and abdominal pain. Both infliximab and adalimumab have been used with success for moderate-to-severe UC refractory to conventional therapy. More recently, golimumab, another anti-TNF antibody, has been added to the treatment armamentarium.

In the multi-centre, double-blind, placebo-controlled PURSUIT trial, patients with moderate-to-severe UC randomized to induction therapy with golimumab (200-100 mg, or 100-50 mg at week 0 and 2) achieved clinical response, clinical remission and mucosal healing more frequent than patients randomized to placebo. In the PURSUIT maintenance trial, patients randomized to golimumab every four weeks (100 or 50 mg) maintained clinical response through week 54 significantly more often than patients randomized to placebo. Data on the use of golimumab in daily clinical practice are unavailable.

The aim of the retrospective Belgian multi-centre BE-SMART trial is to evaluate the mid-term outcome of golimumab in patients with moderate-to-severe colitis. The primary endpoint will be steroid-free golimumab continuation at week 26. Secondary endpoints will include (steroid-free) clinical remission, (steroid-free) clinical response, (steroid-free) mucosal healing, (steroid-free) complete mucosal healing hospitalization-free survival, and colectomy-free survival.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory condition causing continuous mucosal inflammation of the colon, affecting the rectum and a variable extent of the colon in continuity.1 Ulcerative colitis is characterised by a relapsing and remitting course. The aetiology is still unknown, but both genetic and environmental factors seem to be crucial. Ulcerative colitis primarily presents in late adolescence and early adulthood, although the diagnosis may be made at any age. Compared with the general population, the quality of life patients with UC experience is low across all dimensions of health.2;3

When deciding the appropriate treatment strategy for active ulcerative colitis one should consider the activity, distribution and pattern of disease.4 Golimumab has been recently indicated for the treatment of moderately to severely active UC in adult patients who have had an inadequate response to conventional therapy including corticosteroids and 6-mercaptopurine (6-MP) or azathioprine (AZA), or who are intolerant to or have medical contraindications for such therapies.5;6 Besides golimumab, also infliximab and adalimumab are indicated and reimbursed for the treatment of adults with UC.7-9

In the multi-center, double-blind, placebo-controlled PURSUIT trial, patients with established diagnosis of UC and moderate-to-severe disease activity were randomized to receive golimumab 200 mg followed by 100 mg, or 400 mg followed by 200 mg, or twice placebo with 2 weeks apart.5 At week 6, significantly greater proportions of patients in the golimumab 200/100 mg and golimumab 400/200 mg groups (51.8%, and 55.0%, respectively) were in clinical response than patients assigned to placebo (29.7%; P<0.0001 for both comparisons). The efficacy of both golimumab induction regimens was also demonstrated for the major secondary endpoints of clinical remission, mucosal healing, and improvement from baseline in the IBDQ score, all at week 6. In term of safety, similar proportions of patients reported adverse events through week 6 across groups (37.5%, 200/100 mg; 38.9%, 400/200 mg; and 38.2%, placebo).

In a study extension of PURSUIT, patients who responded to induction therapy with golimumab (n=464) were randomly assigned to groups given placebo or injections of 50 or 100 mg golimumab every 4 weeks through week 52.6 Patients who responded to placebo in the induction study continued to receive placebo, while non-responders in the induction study received 100 mg golimumab. The primary endpoint, clinical response maintained through week 54, was observed in 47.1% of patients receiving 50 mg golimumab, 50.6% receiving 100 mg golimumab, and 31.4% receiving placebo (P=0.010 and P<0.001, respectively). At weeks 30 and 54, a higher percentage of patients who received 100 mg golimumab were in clinical remission and had mucosal healing (28.6% and 43.5%) than patients given placebo (15.4% and 26.9%; P=0.003 and P=0.001, respectively) or 50 mg golimumab (23.5% and 41.8%, respectively). Data in daily clinical practice are currently unavailable.

Of note, infliximab requires an intravenous route, and should therefore be administered at the hospital. Altogether, with both transport and monitoring phases, this administration can last more than a half day. In addition, it can be logistically challenging for some patients to reach the hospital (long distance, difficult public transport, significantly altered health condition, …). Subcutaneous therapy can be administered at home and is therefore a very convenient alternative against absenteeism for patients with an active life (workers, students) as well as for patients with challenges in reaching the hospital. In a recent prospective survey in Switzerland, the majority of anti-TNF naïve patients with Crohn's disease preferred subcutaneous administration with either adalimumab (36%) or certolizumab pegol (28%) compared to intravenous infliximab (25%).10 The patients' decision in selecting a specific anti-TNF drug was influenced by ease of use (69%), time required for therapy (34%), time interval between application of the drug (31%), scientific evidence for efficacy (19%), and fear of syringes (10%). Golimumab can therefore be a relevant alternative to infliximab and adalimumab, and can improve these patients' adherence thanks to the lack of either interference with everyday life or hurdles in reaching the hospital, and the need of only one injection every four weeks.

Golimumab currently exists in a prefilled syringe and an auto-injector device (Smartject™). In the recent open-label, multi-centric, prospective GO-MORE study in patients with active rheumatoid arthritis, patients injected 50 mg subcutaneous golimumab once monthly for 6 months. Patients reported use preferences and auto-injector evaluations by questionnaire. Patient auto-injector ratings were favourable overall (e.g. ease of use, pain).11 A similar Belgian trial has been conducted in patients initiating golimumab for moderate-to-severe UC (SMART, ClinicalTrials.gov NCT02155335). In this trial, 100 patients with moderate-to-severe UC, who were either anti-TNF naïve or previously failed infliximab therapy, and previously did not perform self-injection for any indication, have been randomized (1:1) to start crossover therapy with two injections of 50 mg golimumab supplied in a prefilled syringe, and two injections of 50 mg golimumab supplied in an auto-injector device. The efficacy of golimumab therapy will not be evaluated in the SMART study, but this patient population is an ideal cohort to evaluate the short- and mid-term outcome of golimumab monotherapy in real life, and to compare these data with the PURSUIT clinical trial data.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Established diagnosis of UC for at least 3 months
3. Moderate-to-severe ulcerative colitis (Mayo score ≥ 6, including endoscopic sub-score ≥ 2)
4. Previous conventional therapy for a period of at least 3 months with aminosalicylates and at least 3 months with corticosteroids or 6-mercaptopurine (6-MP) or azathioprine (AZA), unless the participant is intolerant to, or has contraindications to these treatments
5. The patients should be

   1. Anti-tumour necrosis factor (anti-TNF) naive participants, OR
   2. Anti-TNF experienced, either not responding, partially responding, or intolerant to treatment with infliximab
6. Sexually active women of child-bearing potential must agree to use a medically accepted method of contraception while receiving study drug and for 6 months after the stop of study drug
7. Willing and able to provide written informed consent

Exclusion Criteria:

1. Has a history of prior self-injection of any agent for any reason
2. Diagnosis of inflammatory bowel disease (IBD) type unclassified or Crohn's disease
3. Previous (procto)colectomy for ulcerative colitis
4. Patients with an ostomy
5. Previous therapy with adalimumab
6. Patients with acute severe IV steroid refractory colitis
7. Concomitant use of other biologic agents
8. Active tuberculosis (TB) within 12 months prior to the first injection or has suspected latent TB as indicated by a positive tuberculin skin test or Interferon gamma (IFNγ) release assay. In case of latent TB, a pneumologist should be contacted and the patient should be treated prophylactically
9. Active clinical non-tuberculous mycobacterial infection or opportunistic infection (e.g. cytomegalovirus, Pneumocystis jiroveci, aspergillosis), within 6 months prior to the first injection
10. Active infection and/or serious infection (e.g. HIV, hepatitis, pneumonia, pyelonephritis, severe sepsis) within 6 months prior to the first study drug administration
11. Live viral or bacterial vaccination within 3 months prior to the first study injection or Bacillus Calmette-Guerin vaccination within 12 months prior to the first study drug injection
12. Evidence of heart failure of New York Heart Association (NYHA) class 3-4
13. History of demyelinating disease such as multiple sclerosis or optic neuritis
14. History of systemic lupus erythematosus
15. History of lymphoproliferative disease, or any unknown malignancy or history of malignancy within the prior 5 years, with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence
16. Active hepatitis B infection
17. Allergy or sensitivity to golimumab or its excipients
18. Pregnant or breast feeding
19. Sensitive to latex
20. Patients with any condition that would prevent completion of the study including history of drug or alcohol abuse, history of mental illness, or history of noncompliance with treatments or visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred patients who participated to the SMART study (EudraCT 2014-000656-29), with moderate-to-severe ulcerative colitis, who are either anti-TNF naïve or who previously failed infliximab therapy, and previously did not perform self-injection for any indication
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Steroid-free clinical response at week 26 | Week 26
  Percentage of participants with steroid-free clinical response at week 26 Clinical response was defined as a decrease from baseline in the total Mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the sub-score for rectal bleeding of at least 1 point or an absolute sub-score for rectal bleeding of 0 or 1

SECONDARY OUTCOMES:
Golimumab continuation at week 26 | Week 26
  Percentage of participants who are still receiving golimumab at week 26 and are free of steroids and did not require treatment optimization with golimumab
(Steroid-free) Clinical remission at week 14 | Week 14
  Percentage of patients who achieved (steroid-free) clinical remission at week 12-14 Clinical remission is defined as a total Mayo score of 2 points or lower, with no individual sub-score exceeding 1 point
(Steroid-free) Clinical remission at week 26 | Week 26
  Percentage of patients who achieved (steroid-free) clinical remission at week 26 Clinical remission is defined as a total Mayo score of 2 points or lower, with no individual sub-score exceeding 1 point
(Steroid-free) Clinical remission at week 52 | Week 52
  Percentage of patients who achieved (steroid-free) clinical remission at week 48-52 Clinical remission is defined as a total Mayo score of 2 points or lower, with no individual sub-score exceeding 1 point
(Steroid-free) Clinical response at week 14 | Week 14
  Percentage of patients who achieved (steroid-free) clinical response at week 12-14 Clinical response was defined as a decrease from baseline in the total Mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the sub-score for rectal bleeding of at least 1 point or an absolute sub-score for rectal bleeding of 0 or 1
(Steroid-free) Clinical response at week 52 | Week 52
  Percentage of patients who achieved (steroid-free) clinical response at week 48-52 Clinical response was defined as a decrease from baseline in the total Mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the sub-score for rectal bleeding of at least 1 point or an absolute sub-score for rectal bleeding of 0 or 1
(Steroid-free) mucosal healing at week 14 | Week 14
  Percentage of patients who achieved (steroid-free) mucosal healing at week 12-14 Mucosal healing is defined as an absolute sub-score for endoscopy of 0 or 1, and will only be evaluated in patients with an endoscopy sub-score of 2 or 3 at baseline
(Steroid-free) mucosal healing at week 52 | Week 52
  Percentage of patients who achieved (steroid-free) mucosal healing at week 48-52 Mucosal healing is defined as an absolute sub-score for endoscopy of 0 or 1, and will only be evaluated in patients with an endoscopy sub-score of 2 or 3 at baseline
(Steroid-free) complete mucosal healing at week 14 | Week 14
  Percentage of patients who achieved (steroid-free) complete mucosal healing at week 12-14 Complete mucosal healing is defined as an absolute sub-score for endoscopy of 0, and will only be evaluated in patients with an endoscopy sub-score of 2 or 3 at baseline
(Steroid-free) complete mucosal healing at week 52 | Week 52
  Percentage of patients who achieved (steroid-free) complete mucosal healing at week 48-52 Complete mucosal healing is defined as an absolute sub-score for endoscopy of 0, and will only be evaluated in patients with an endoscopy sub-score of 2 or 3 at baseline
Sustained clinical remission | Week 52
  Percentage of patients who achieved sustained clinical remission with clinical remission at weeks 12-14, week 26, and week 48-52.
Sustained clinical response | Week 52
  Percentage of patients who achieved sustained clinical response with clinical response at weeks 12-14, week 26, and week 48-52.
Need for colectomy by week 52 | Week 52
  Percentage of patients requiring colectomy within 52 weeks
Need for UC related hospitalization by week 52 | Week 52
  Percentage of patients requiring hospitalization for UC within 52 weeks
Golimumab discontinuation-free survival | Week 52
  Percentage of patients still under golimumab at week 52
Golimumab related (serious) adverse events | Week 52
  Percentage of patients developing (serious) adverse events under golimumab therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: Undecided